CLINICAL TRIAL: NCT06127849
Title: A Randomized, Placebo-controlled, Blinded Study to Evaluate Efficacy of EB-PA as Protein Amplifier for Skeletal Muscle Strength & Growth
Brief Title: A Study to Evaluate Efficacy of EB-PA as Protein Amplifier for Skeletal Muscle Strength & Growth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: EB/230701/EB-PA/SMSG
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Skeletal Muscle Strength & Growth
MeSH Terms: interventions — Resistance Training; Capsules; Whey Proteins

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blinded study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resistance Training + Placebo (Capsule) + Placebo (Sachet) (Placebo Comparator): A sachet of 20 gms of Placebo dissolved in 200-300 ml water. One sachet to be taken in the Morning and one in the evening.
  One capsule of placebo to be taken 30 minutes after placebo sachet in the morning.
  Interventions: Dietary Supplement: Resistance Training + Placebo (Capsule) + Placebo (Sachet)
- Resistance Training + Whey protein (40 gms) + Placebo (Capsule) (Active Comparator): A sachet of 20 gms of Whey protein isolate (WPI) dissolved in 200-300 ml water. One sachet to be taken in the Morning and one in the evening.
  One capsule of Placebo to be taken 30 minutes after whey protein in the morning.
  Interventions: Dietary Supplement: Resistance Training + Whey protein (40 gms) + Placebo (Capsule)
- Resistance Training + Whey protein (40 gms) + EB-PA (500 mg) (Active Comparator): A sachet of 20 gms of Whey protein isolate (WPI) dissolved in 200-300 ml water. One sachet to be taken in the Morning and one in the evening.
  One capsule of EB0-PA to be taken 30 minutes after whey protein in the morning.
  Interventions: Dietary Supplement: Resistance Training + Whey protein (40 gms) + EB-PA (500 mg)

INTERVENTIONS:
Dietary Supplement: Resistance Training + Placebo (Capsule) + Placebo (Sachet) — * Placebo sachet of 20 gms dissolved in 200-300 ml water. One sachet to be taken in the Morning and one in the evening.
  * One Placebo capsule to be taken 30 minutes after sachet in the morning.
  Arms: Resistance Training + Placebo (Capsule) + Placebo (Sachet)
Dietary Supplement: Resistance Training + Whey protein (40 gms) + Placebo (Capsule) — A sachet of 20 gms of Whey protein isolate (WPI) dissolved in 200-300 ml water. One sachet to be taken in the Morning and one in the evening.
  - One Placebo capsule to be taken 30 minutes after whey protein in the morning
  Arms: Resistance Training + Whey protein (40 gms) + Placebo (Capsule)
Dietary Supplement: Resistance Training + Whey protein (40 gms) + EB-PA (500 mg) — * A sachet of 20 gms of Whey protein isolate (WPI) dissolved in 200-300 ml water. One sachet to be taken in the Morning and one in the evening.
  * One capsule of EB-PA to be taken 30 minutes after whey protein in the morning
  Arms: Resistance Training + Whey protein (40 gms) + EB-PA (500 mg)

SUMMARY:
The present study is a randomized, placebo-controlled, double blinded study to evaluate efficacy of EB-PA as protein amplifier for skeletal muscle strength & growth in males with active lifestyle. Approximately 160 subjects aged between ≥ 20 and ≤ 35 years will be screened and 138 participants are to be randomized. Both the IP and placebo study arms will have at least 40 completed subjects after accounting for the screening failure and dropout/withdrawal rate of 14% and 13 % respectively (Total 120 completers). The treatment duration for all the study subjects will be 30 days. The sustained effect of the product will be observed for next 7 days, wherein, the subjects will be abstaining from the protein and IP supplementation and will exercise at their ease.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 20 - 35 years with active lifestyle with moderate physical activity level as per International Physical Activity Questionnaire.
* Recreationally gym goer with history of at least 1 month of endurance training (E.g.: functional exercises)
* Not participating in resistance type training (E.g.: external or body weight training) for ≥3 months prior to screening.
* Body mass index (BMI) 22 - 29.9 kg/ m2.
* Individuals with a 1-RM strength defined by Upper Body ≥ 25 Kgs and Lower Body ≥ 100 Kgs will be included in the study.
* Ready to refrain from caffeinated products and intense strength/ endurance exercise for 24 hrs prior to the exercise lab visit.
* Fasting Blood Glucose ≤ 110 mg/ dl.
* Systolic Blood Pressure ≤ 129 mmHg and Diastolic Blood Pressure ≤ 89 mmHg.
* TSH (thyroid stimulating hormone) ≥ 0.4 and ≤ 4.9 mIU/L.

Exclusion Criteria:

* Engaged in structured weight training for more than 3 months prior to screening.
* Presence of chronic disease.
* Changes in body weight more than 4.5 kg (10 pounds) in the past three months as assessed by history.
* Subjects diagnosed with hypertension.
* Subjects who are diagnosed with Type I Diabetes Mellitus and Type II Diabetes Mellitus.
* History or presence of clinically significant renal, hepatic, endocrine, biliary, gastrointestinal, pancreatic or neurologic disorders.
* Allergy to whey protein or herbal ingredients.
* Subjects who have any other disease or condition, or are using any medication, that in the judgment of the investigator would put them at unacceptable risk for participation in the study or may interfere with evaluations in the study or noncompliance with treatment or visits.
* Subjects who have been part of a clinical study within 90 days prior to the screening.
* Subjects who have used whey or other supplemental proteins anytime in last 3 months.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 138 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-06-05 (Estimated)

PRIMARY OUTCOMES:
To assess improvement in muscle strength after administration of Investigational Product (IP) as assessed by increase in lower body 1 RM (repetition maximum) weight from baseline. | Day 30
  The maximum weight that can be lifted once with the correct lifting technique is known as the 1-RM. The 1-RM will be determined by the Brzycki equation using calculator as follows: Weight ÷ [1.0278 - (0.0278 × Number of repetitions)].
To assess improvement in muscle strength after administration of Investigational Product (IP) as assessed by increase in upper body 1 RM (repetition maximum) weight from baseline. | Day 30
  The maximum weight that can be lifted once with the correct lifting technique is known as the 1-RM. The 1-RM will be determined by the Brzycki equation using calculator as follows: Weight ÷ [1.0278 - (0.0278 × Number of repetitions)].

SECONDARY OUTCOMES:
To assess the effect of Investigational Product (IP) on Increase in muscle endurance as assessed by increase in exercise volume calculated as load x number of repetition (upper + lower body exercise) completed at ≥70% of screening 1-RM. | Day 0 to Day 30
  The maximum weight that can be lifted once with the correct lifting technique is known as the 1-RM. The 1-RM will be determined by the Brzycki equation using calculator as follows: Weight ÷ [1.0278 - (0.0278 × Number of repetitions)].
To assess the effect of Investigational Product (IP) on Increase in muscle (hamstring) flexibility as assessed by increase in distance for V sit & reach test. | Day 0 to Day 30
  V sit and reach test is performed to measure the flexibility of the lower back and back thigh muscles.
To assess the effect of IP on improvement in muscle mass as indicated by increase in fat free mass (FFM), lean muscle mass and android fat by DXA. | Day 0 to Day 30
  Total body scans will be performed using a device with its scan mode already determined automatically by the device operating system within the manufacture specification.
To assess the effect of IP on improvement in grip strength as indicated by increase in non-dominant hand grip strength. | Day 0 to Day 30
  Each subject will perform the test three times approximately with 25±5 sec relaxations between the session. The participant should be instructed to squeeze the dynamometer until the grip is stable. For 3 sets, the reading will be noted in Kg and an average of 3 readings will be calculated.
To assess the effect of IP on Improvement in metabolic health as indicated by waist to height ratio. | Day 0 to Day 30
  Waist circumference (WC) will be measured at the end of a normal expiration using a non-stretchable measuring tape.
To assess the sustained effect of IP on muscle strength as assessed by Maintenance of lower body 1 RM weight | Day 30 To 37
  The maximum weight that can be lifted once with the correct lifting technique is known as the 1-RM. The 1-RM will be determined by the Brzycki equation using calculator as follows: Weight ÷ [1.0278 - (0.0278 × Number of repetitions)].
To assess the sustained effect of IP on muscle strength as assessed by Maintenance of upper body 1RM weight | Day 30 To 37
  The maximum weight that can be lifted once with the correct lifting technique is known as the 1-RM. The 1-RM will be determined by the Brzycki equation using calculator as follows: Weight ÷ [1.0278 - (0.0278 × Number of repetitions)].

CONTACTS AND LOCATIONS:
Locations (3):
- India (3):
  - Dr. Khare's Clinic, Mumbai, Maharashtra
  - Nirmala Clinic, Mumbai, Maharashtra
  - Dr. Preeti Bawaskar's Clinic, Thane, Maharashtra

IPD SHARING:
Plan to Share IPD: Undecided